CLINICAL TRIAL: NCT03872947
Title: A Phase 1b, Multicenter Study to Determine the Dose, Safety, Efficacy and Pharmacokinetics of TRK-950 When Used in Combinations With Selected Anti-Cancer Treatment Regimens in Patients With Selected Advanced Solid Tumors
Brief Title: A Study of TRK-950 in Combinations With Anti-Cancer Treatment Regimens in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 950P1V02
Record Dates: First submitted 2019-03-07; First posted 2019-03-13 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor; Colorectal Cancer; Cholangiocarcinoma; Bladder Cancer; Ovarian Cancer; Gastric Cancer; Palpable Subcutaneous Malignant Lesions; Renal Cell Carcinoma; Melanoma; Epithelial Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Cholangiocarcinoma; Urinary Bladder Neoplasms; Ovarian Neoplasms; Stomach Neoplasms; Carcinoma, Renal Cell; Melanoma; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Irinotecan; Leucovorin; Fluorouracil; Gemcitabine; Cisplatin; Carboplatin; Ramucirumab; Paclitaxel; Nivolumab; pembrolizumab; Bevacizumab; 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (15):
- Arm A: TRK-950 + FOLFIRI (Experimental): * Colorectal Cancer
  * TRK-950 will be administered intravenously (IV) on days 1, 8, 15, and 22 of a 28-day cycle. On days 1 and 15 Irinotecan will be administered IV. Leucovorin will be infused to match the duration of the irinotecan infusion. 5-FU will be administered as IV bolus, followed by TRK-950 administration. After the TRK-950, 5-FU will be administered by a continuous infusion.
  Interventions: Biological: TRK-950; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU
- Arm B: TRK-950 + Gemcitabine/Cisplatin (Experimental): * Cholangiocarcinoma or Bladder Cancer
  * TRK-950 will be administered IV on days 1, 8 and 15 of a 21-day cycle. After the administration of TRK-950 on days 1 and 8, Cisplatin will be administered by infusion. Then, Gemcitabine will be administered as an IV infusion.
  Interventions: Biological: TRK-950; Drug: Gemcitabine; Drug: Cisplatin
- Arm C: TRK-950 + Gemcitabine/Carboplatin (Experimental): * Ovarian Cancer
  * TRK-950 will be administered IV on days 1, 8 and 15 of a 21-day cycle. After the administration of TRK-950 on days 1 and 8, Gemcitabine will be administered as an intravenous infusion. On day 1, following the administration of TRK-950 and Gemcitabine, Carboplatin will be administered IV.
  Interventions: Biological: TRK-950; Drug: Gemcitabine; Drug: Carboplatin
- Arm D: TRK-950 + Ramucirumab/Paclitaxel (Experimental): * Gastric Cancer
  * TRK-950 will be administered IV on days 1, 8, 15, and 22 of a 28-day cycle. After the administration of TRK-950 on days 1 and 15, Ramucirumab will be administered as an IV infusion. Paclitaxel will be dosed on days 1, 8 and 15, after the Ramucirumab on days 1 and 15 and after the TRK-950 on day 8.
  Interventions: Biological: TRK-950; Drug: Ramucirumab; Drug: Paclitaxel
- Arm E: TRK-950 + PD1 inhibitors (Experimental): •Solid Tumors
  E-1: TRK-950 + Nivolumab
  •TRK-950 will be administered IV on days 1, 8, 15, and 22 of a 28-day cycle. After the administration of TRK-950 on days 1 and 15, Nivolumab will be administered as an IV infusion.
  E-2: TRK-950 + Pembrolizumab
  •TRK-950 will be administered IV on days 1, 8 and 15 of a 21-day cycle. After the administration of TRK-950 on day 1, Pembrolizumab will be administered as an IV infusion.
  Interventions: Biological: TRK-950; Drug: Nivolumab; Drug: Pembrolizumab
- Arm F: TRK-950 + Imiquimod Cream (Experimental): * Palpable subcutaneous malignant lesions
  * TRK-950 will be administered IV on days 1, 8 and 15 of a 21-day cycle. Imiquimod cream is to be applied 5 of 7 days in a row with 2 days rest for a maximum of 2 cycles (total 6 weeks).
  Interventions: Biological: TRK-950; Drug: Imiquimod Cream
- Arm G: TRK-950 + Bevacizumab (Experimental): * Renal Cell Carcinoma
  * TRK-950 will be administered IV on days 1, 8, 15, and 22 of a 28-day cycle. After the administration of TRK-950 on days 1 and 15, Bevacizumab will be administered as an IV infusion.
  Interventions: Biological: TRK-950; Drug: Bevacizumab
- Arm H: TRK-950 + PD1 inhibitors (Experimental): •Melanoma
  H-1: TRK-950 + Nivolumab
  •TRK-950 will be administered IV on days 1, 8, 15, and 22 of a 28-day cycle. After the administration of TRK-950 on days 1 and 15, Nivolumab will be administered as an IV infusion.
  H-2: TRK-950 + Pembrolizumab
  •TRK-950 will be administered IV on days 1, 8 and 15 of a 21-day cycle. After the administration of TRK-950 on day 1, Pembrolizumab will be administered as an IV infusion.
  Interventions: Biological: TRK-950; Drug: Nivolumab; Drug: Pembrolizumab
- Arm J: TRK-950 + FOLFIRI (Experimental): * Colorectal Cancer
  * TRK-950 will be administered IV on days 1, 8, 15, and 22 of a 28-day cycle. On days 1 and 15 Irinotecan will be administered IV. Leucovorin will be infused to match the duration of the irinotecan infusion. 5-FU will be administered as IV bolus, followed by TRK-950 administration. After the TRK-950, 5-FU will be administered by a continuous infusion.
  Interventions: Biological: TRK-950; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU
- Arm K: TRK-950 + Gemcitabine / Carboplatin / Bevacizumab (Experimental): * Platinum Sensitive epithelial ovarian, primary peritoneal or fallopian tube cancer
  * TRK-950 will be administered IV on days 1, 8 and 15 of a 21-day cycle. On all dosing days, TRK-950 will be administered IV after the relevant combination regimen is dosed. Gemcitabine will be administered as an intravenous infusion on days 1 and 8. On day 1, following the administration of Gemcitabine, Carboplatin will be administered as an intravenous infusion. Also on Day 1 of each cycle, Bevacizumab will be administered IV next. After 6 cycles of chemotherapy the patient will be transitioned to maintenance treatment. On Day 1 of each maintenance cycle, Bevacizumab will be administered IV. Maintenance treatment will be continued as long as there is no evidence of progressive disease.
  Interventions: Biological: TRK-950; Drug: Gemcitabine; Drug: Carboplatin; Drug: Bevacizumab
- Arm O: TRK-950 + PLD (Experimental): * Platinum Resistant epithelial ovarian, primary peritoneal or fallopian tube cancer
  * TRK-950 will be administered IV on days 1, 8, 15, and 22 of a 28-day cycle. PLD will be dosed as IV on Day 1 of each cycle. On days that TRK-950 and PLD are both dosed, PLD will be dosed first.
  Interventions: Biological: TRK-950; Drug: PLD
- Arm Q: TRK-950 + Ramucirumab/Paclitaxel (Experimental): * Gastric cancer
  * TRK-950 will be administered IV on days 1, 8, 15, and 22 of a 28-day cycle. On all dosing days, TRK-950 will be administered IV after the relevant combination regimen is dosed. On days 1 and 15, ramucirumab will be administered IV. Paclitaxel will be dosed on days 1, 8 and 15, after ramucirumab on days 1 and 15, before TRK-950 on day 8.
  Interventions: Biological: TRK-950; Drug: Ramucirumab; Drug: Paclitaxel
- Arm R: TRK-950 + Bevacizumab (Experimental): * Renal cell carcinoma cancer
  * TRK-950 will be administered IV on days 1, 8, 15, and 22 of a 28-day cycle. Bevacizumab will be dosed as IV on Day 1 and 15 of each cycle. On days that TRK-950 and Bevacizumab are both dosed, Bevacizumab will be dosed first.
  Interventions: Biological: TRK-950; Drug: Bevacizumab
- Arm S: TRK-950 + Carboplatin / PLD/ Bevacizumab (Experimental): * Platinum Sensitive epithelial ovarian, primary peritoneal or fallopian tube cancer
  * Treatment Phase: TRK-950 will be administered IV on days 1 and 15 of a 28-day cycle. Carboplatin will be administered as an intravenous infusion on day 1. On day 1, following the administration of Carboplatin, PLD will be administered as an intravenous infusion. Also on Day 1 of each cycle, Bevacizumab will be administered IV next.
  On days 1 and 15, TRK-950 will be administered IV after the Bevacizumab infusion.
  • Maintenance Phase: After 6 cycles of chemotherapy, the patient will be transitioned to maintenance treatment. On Day 1 of each maintenance cycle, Bevacizumab will be administered IV. Following the Bevacizumab administration, TRK-950 will be administered IV. Maintenance treatment will be continued as long as there is no evidence of progressive disease.
  Interventions: Biological: TRK-950; Drug: Carboplatin; Drug: Bevacizumab; Drug: PLD
- Arm T: TRK-950 + Paclitaxel (Experimental): * Platinum Resistant epithelial ovarian, primary peritoneal or fallopian tube cancer
  * TRK-950 will be administered IV on days 1, 8, 15, and 22 of a 28-day cycle. On days 1, 8 and 15 of each cycle, Paclitaxel will be dosed on IV
  Interventions: Biological: TRK-950; Drug: Paclitaxel

INTERVENTIONS:
Biological: TRK-950 — 10 mg/kg administered intravenously over 60 minutes (weekly)
  Arms: Arm A: TRK-950 + FOLFIRI; Arm B: TRK-950 + Gemcitabine/Cisplatin; Arm C: TRK-950 + Gemcitabine/Carboplatin; Arm D: TRK-950 + Ramucirumab/Paclitaxel; Arm E: TRK-950 + PD1 inhibitors; Arm F: TRK-950 + Imiquimod Cream; Arm G: TRK-950 + Bevacizumab; Arm H: TRK-950 + PD1 inhibitors; Arm J: TRK-950 + FOLFIRI; Arm T: TRK-950 + Paclitaxel
Biological: TRK-950 — 5 mg/kg administered intravenously over 60 minutes (weekly)
  Arms: Arm K: TRK-950 + Gemcitabine / Carboplatin / Bevacizumab; Arm O: TRK-950 + PLD; Arm Q: TRK-950 + Ramucirumab/Paclitaxel; Arm R: TRK-950 + Bevacizumab
Biological: TRK-950 — Treatment Phase: 20 mg/kg administered intravenously over 60 minutes (bi-weekly) Maintenance Phase: 30 mg/kg administered intravenously over 60 minutes (every 3 weeks)
  Arms: Arm S: TRK-950 + Carboplatin / PLD/ Bevacizumab
Drug: Irinotecan — Intravenously over 30 - 90 minutes
  Arms: Arm A: TRK-950 + FOLFIRI; Arm J: TRK-950 + FOLFIRI
Drug: Leucovorin — Intravenously over 30 - 90 minutes
  Arms: Arm A: TRK-950 + FOLFIRI; Arm J: TRK-950 + FOLFIRI
Drug: 5-FU — Intravenously bolus and intravenously for two days
  Arms: Arm A: TRK-950 + FOLFIRI; Arm J: TRK-950 + FOLFIRI
Drug: Gemcitabine — Intravenously over 30 minutes
  Arms: Arm B: TRK-950 + Gemcitabine/Cisplatin; Arm C: TRK-950 + Gemcitabine/Carboplatin; Arm K: TRK-950 + Gemcitabine / Carboplatin / Bevacizumab
Drug: Cisplatin — Intravenously over 60 minutes
  Arms: Arm B: TRK-950 + Gemcitabine/Cisplatin
Drug: Carboplatin — Intravenously per package insert
  Arms: Arm C: TRK-950 + Gemcitabine/Carboplatin; Arm K: TRK-950 + Gemcitabine / Carboplatin / Bevacizumab; Arm S: TRK-950 + Carboplatin / PLD/ Bevacizumab
Drug: Ramucirumab — Intravenously over 60 minutes
  Arms: Arm D: TRK-950 + Ramucirumab/Paclitaxel; Arm Q: TRK-950 + Ramucirumab/Paclitaxel
Drug: Paclitaxel — Intravenously
  Arms: Arm D: TRK-950 + Ramucirumab/Paclitaxel; Arm Q: TRK-950 + Ramucirumab/Paclitaxel; Arm T: TRK-950 + Paclitaxel
Drug: Nivolumab — Intravenously over 30 minutes
  Arms: Arm E: TRK-950 + PD1 inhibitors; Arm H: TRK-950 + PD1 inhibitors
Drug: Pembrolizumab — Intravenously over 30 minutes
  Arms: Arm E: TRK-950 + PD1 inhibitors; Arm H: TRK-950 + PD1 inhibitors
Drug: Imiquimod Cream — Topically
  Arms: Arm F: TRK-950 + Imiquimod Cream
Drug: Bevacizumab — Intravenously over 90 minutes for the first dose, over 60 for the second dose and over 30 minutes for all subsequent doses
  Arms: Arm G: TRK-950 + Bevacizumab; Arm K: TRK-950 + Gemcitabine / Carboplatin / Bevacizumab; Arm R: TRK-950 + Bevacizumab; Arm S: TRK-950 + Carboplatin / PLD/ Bevacizumab
Drug: PLD — Intravenously over 60 minutes
  Arms: Arm O: TRK-950 + PLD; Arm S: TRK-950 + Carboplatin / PLD/ Bevacizumab

SUMMARY:
The main purpose of this study is to establish the safety and the recommended dose of TRK-950 in combination with FOLFIRI, Gemcitabine / Cisplatin, Gemcitabine / Carboplatin, Ramucirumab / Paclitaxel, PD1 inhibitors (Nivolumab or Pembrolizumab), and Imiquimod Cream, Bevacizumab, Gemcitabine / Carboplatin / Bevacizumab, Pegylated liposomal doxorubicin (PLD), Carboplatin / PLD / Bevacizumab and Paclitaxel for selected advanced solid tumors.

DETAILED DESCRIPTION:
This study is an open-label, Phase 1b study evaluating TRK-950 in combination with 1) FOLFIRI or 2) Gemcitabine / Cisplatin or 3) Gemcitabine / Carboplatin or 4) Ramucirumab/Paclitaxel or 5) PD1 inhibitors (Nivolumab or Pembrolizumab) or 6) Imiquimod Cream for subcutaneous lesions 7) Bevacizumab 8) Gemcitabine / Carboplatin / Bevacizumab, 9)PLD, 10) Carboplatin / PLD / Bevacizumab or 11) Paclitaxel in Patients with Selected Advanced Solid Tumors. The objectives of this study are to determine the safety, tolerability, MTD, recommended Phase 2 dose (RP2D), PK, and preliminary anti-tumor activity of TRK-950 when used in combination with other treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid malignancy for which the following treatment regimens are warranted:
* Arm A. Colorectal Cancer with no prior history of treatment with Irinotecan alone or in combination: FOLFIRI as standard of care
* Arm B. Cholangiocarcinoma, Bladder Cancer with no prior history of treatment with Gemcitabine alone or in combination: Gemcitabine / Cisplatin as standard of care
* Arm C. Ovarian Cancer who have relapsed at least 6 or more months after completion of a previous platinum-based therapy and have no prior history of treatment with gemcitabine alone or in combination: Gemcitabine / Carboplatin as standard of care
* Arm D. Gastric Cancer including Gastroesophageal Junction with no prior history of treatment with Ramucirumab, Paclitaxel or any Taxane class drug: Ramucirumab / Paclitaxel as standard of care
* Arm E. Solid Tumors: Eligible for PD1 Inhibitor (Nivolumab or Pembrolizumab) monotherapy as standard of care according to the approved drug label by the relevant regulatory authority
* Arm F. Locally advanced or metastatic disease in a cancer with at least one palpable subcutaneous malignant lesion (≤ 2 cm in diameter) for treatment with TRK-950 and Imiquimod cream (US Sites Only)
* Arm G. Renal Cell Carcinoma with no prior history of treatment with Bevacizumab alone or in combination: Bevacizumab for use in a fourth line or later treatment
* Arm H. Melanoma patients who progressed while taking Nivolumab, Pembrolizumab, or Ipilimumab, within the last 6 months prior to cycle 1 day 1
* Arm J. Colorectal Cancer patients who progressed on FOLFIRI or any other Irinotecan-containing therapy regimen within the last 6 months prior to cycle 1 day 1
* Arm K. (US Sites Only). Platinum Sensitive epithelial ovarian, primary peritoneal or fallopian tube cancer with ≤ 2 prior treatment lines who have recurred > 6 months after most recent platinum-based chemotherapy and who are eligible for gemcitabine, carboplatin, and Bevacizumab as standard of care for dosing of TRK-950
* Arm O. Platinum Resistant epithelial ovarian, primary peritoneal or fallopian tube cancer with ≤ 5 prior treatment regimens, as defined below and who are eligible for topotecan or pegylated liposomal doxorubicin as standard of care for dosing of TRK-950

  * Patients who have only had 1 line of platinum-based therapy must have received at least 4 cycles of platinum, must have had a response, and then progressed between 3 months and less than or equal to 6 months after the last date of platinum.
  * Patients who have received 2 to 5 lines of prior therapy must have received at least 4 cycles of platinum and then progressed within 6 months after the date of the last dose of platinum.
  * Prior treatment with bevacizumab is required for patients with 1 to 2 prior lines of therapy
* Arm Q. Gastric Cancer including GEJ cancer with only 1 prior treatment regimen, which recurred during or within 4 months after frontline treatment, and no prior history of treatment with Ramucirumab, Paclitaxel or any Taxane class drug for metastatic disease: eligible to receive Ramucirumab/Paclitaxel as standard of care
* Arm R. Clear cell renal cell carcinoma with no prior history of treatment with Bevacizumab alone or in combination: Bevacizumab for use in a fourth line or later treatment.
* Arm S. Platinum Sensitive epithelial ovarian, primary peritoneal or fallopian tube cancer with ≤ 2 prior treatment lines who have recurred > 182 days after most recent platinum-based chemotherapy and who are eligible for carboplatin, PLD, and bevacizumab as standard of care

  * The histological subtypes of the carcinoma that qualify for enrollment include serous adenocarcinoma, endometrioid adenocarcinoma, carcinosarcoma of the ovary, or adenocarcinoma not otherwise specified (NOS)
  * Patients with or without the breast cancer susceptibility 1/2 (BRCA1/2) mutations are eligible, provided that patients with the BRCA1/2 mutations have previously received PARP inhibitor treatment
* Arm T. Platinum Resistant epithelial ovarian, primary peritoneal or fallopian tube cancer with ≤ 5 prior treatment regimens, or as defined below, and who are eligible for paclitaxel as standard of care

  * Patients who have only had 1 line of platinum-based therapy must have received at least 4 cycles of platinum, must have had a response (complete response/remission (CR) or partial response/remission (PR), and then progressed between 90 days to less than 183 days after the last date of platinum.
  * Patients who have received multiple lines of platinum therapy must have progressed on the latest platinum, or within 183 days after the date of the last dose of the latest platinum
  * Patients with or without the BRCA1/2 mutations are eligible, provided that patients with the BRCA1/2 mutations have previously received PARP inhibitor treatment
  * Prior treatment with bevacizumab is required for patients with 1 to 2 prior lines of therapy
  * The histological subtypes of the carcinoma that qualify for enrollment include serous adenocarcinoma, endometrioid adenocarcinoma, carcinosarcoma of the ovary, or adenocarcinoma not otherwise specified (NOS)
* Primary or metastatic tumors measurable per RECIST v1.1 on CT scan or by calipers (subcutaneous lesions)
* Karnofsky performance of ≥70
* Life expectancy of at least 3 months
* Age ≥ 18 years
* Signed, written IRB-approved informed consent

Exclusion Criteria:

* Laboratory values or medications that are contraindicated in the selected standard of care treatment regimens
* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy. Prophylactic antibiotics are acceptable.
* Pregnant or nursing women
* Treatment with radiation therapy within 2 weeks, or treatment with surgery, chemotherapy, immunotherapy, targeted therapy or investigational therapy within four weeks prior to initiation of study treatment (6 weeks for nitrosoureas or mitomycin C, and 2 weeks or 5 half-lives whichever is longer for TKIs).
* Unwillingness or inability to comply with procedures required in this protocol
* Known active infection with HIV, hepatitis B, hepatitis C
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Patients who are currently receiving any other investigational agent
* Any contraindicated condition or drug which would make the patient ineligible for the respective treatment regimen that is to be used in combination with TRK-950 (for example, autoimmune disorders for nivolumab or pembrolizumab treatment) as described in the Full Prescribing Information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of patients experiencing treatment emergent adverse events as assessed by CTCAE v5.0 | through study completion, an average of 1 year
Frequency of patients experiencing adverse events of special interest (AESIs) | through study completion, an average of 1 year
Blood pressure | through study completion, an average of 1 year
  mmHg
Heart rate | through study completion, an average of 1 year
  bpm
Respiratory rate | through study completion, an average of 1 year
  bpm
Temperature | through study completion, an average of 1 year
  °F or °C
Weight | through study completion, an average of 1 year
  lbs/kg
Height | through study completion, an average of 1 year
  inches/cm
Performance status using Karnofsky performance status criteria | through study completion, an average of 1 year
QTc interval determined from 12-lead Electrocardiogram | through study completion, an average of 1 year
  msec
QRS interval determined from 12-lead Electrocardiogram | through study completion, an average of 1 year
  msec
Frequency of patients with laboratory abnormalities (Complete Blood Count, Coagulation, Urinalysis and Serum Chemistry) | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Overall response rate (ORR) | through study completion, an average of 1 year
Disease Control Rate (DCR) | through study completion, an average of 1 year
Serum concentration of TRK-950 | through study completion, an average of 1 year
Plasma concentration of Gemcitabine for the first six patients in Arm K | At the beginning of Cycle 1 and Cycle 4 (each cycle is 21 days)
Plasma concentration of Carboplatin for the first six patients in Arm K | At the beginning of Cycle 1 and Cycle 4 (each cycle is 21 days)
Serum concentration of Bevacizumab for the first six patients in Arm K | At the beginning of Cycle 1, Cycle 2, Cycle 4 and Cycle 5 (each cycle is 21 days)
Plasma concentration of PLD for the first six patients in Arm O | At the beginning and middle of Cycle 1 and Cycle 3 (each cycle is 28 days)
Serum concentration of Ramucirumab for the first six patients in Arm Q | At the beginning and middle of Cycle 1 and Cycle 4 (each cycle is 28 days)
Plasma concentration of Paclitaxel for the first six patients in Arm Q | At the beginning of Cycle 1 and Cycle 4 (each cycle is 28 days)
Serum concentration of Bevacizumab for the first six patients in Arm R | At the beginning and middle of Cycle 1 and Cycle 4 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - AOA-HOPE, Tucson, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - HOAG Memorial Hospital Presbyterian, Newport, California
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Atlantic Health System, Morristown, New Jersey
  - Perlmutter Cancer Center at NYU Langone, New York, New York
  - Oncology Associates of Oregon, P.C.(Willamette Valley Cancer Institute and Research Center), Eugene, Oregon
  - Northwest Cancer Specialists, Portland, Oregon
  - Texas Oncology, P.A. Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Downtown Fort Worth Cancer Center, Fort Worth, Texas
  - Virginia Cancer Specialists, PC, Leesburg, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okano F, Saito T, Minamida Y, Kobayashi S, Ido T, Miyauchi Y, Wasai U, Akazawa D, Kume M, Ishibashi M, Jiang K, Aicher A, Heeschen C, Yonehara T. Identification of Membrane-expressed CAPRIN-1 as a Novel and Universal Cancer Target, and Generation of a Therapeutic Anti-CAPRIN-1 Antibody TRK-950. Cancer Res Commun. 2023 Apr 18;3(4):640-658. doi: 10.1158/2767-9764.CRC-22-0310. eCollection 2023 Apr. PMID 37082579